CLINICAL TRIAL: NCT06355206
Title: Natural Course and Therapeutic Effect of Recurrent Acute Pancreatitis: a Prospective Cohort Study
Brief Title: Natural Course and Therapeutic Effect of Recurrent Acute Pancreatitis
Acronym: NACRE
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: NACRE20230306
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cohort Study; Recurrent Acute Pancreatitis
Keywords: recurrent acute pancreatitis; natural course; therapeutic effect
MeSH Terms: conditions — Pancreatitis | interventions — Surgical Procedures, Operative; Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Feces and blood samples from RAP patients will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- recurrent acute pancreatitis: Recurrent acute pancreatitis is generally defined as a condition in which at least two well documented episodes of acute pancreatitis have occurred, with resolution of symptoms between each episode, and absence of morphological criteria for chronic pancreatitis.
  Interventions: Combination Product: endoscopic intervention, surgery or conservative treatment

INTERVENTIONS:
Combination Product: endoscopic intervention, surgery or conservative treatment — Personal information and treatment of the enrolled subjects will be collected.

SUMMARY:
The goal of this observational cohort study is to learn about the etiology, natural course, therapeutic effect and outcome of recurrent acute pancreatitis patients. The main question it aims to answer is:

Does endoscopic intervention, surgery or conservative treatment reduce the recurrence of acute pancreatitis? What are the risk factors affecting the recurrence of acute pancreatitis?

Patients will be closely followed and clinical information will be recorded.

DETAILED DESCRIPTION:
Acute pancreatitis is one of the most common causes of acute hospital admission, which is unpredictable and contributes to high health-care costs even death. Recurrent acute pancreatitis is defined as two or more discrete episodes of acute pancreatitis, and has an estimated annual incidence of 8-10 per 100 000. Cholelithiasis, alcohol and Hyperglyceremia are the most commonly recognized causes of acute pancreatitis. About 80% of RAP patients can be identified through routine investigations identify (include proper history, physical examination, CT, MRI, endoscopic ultrasound); however, in up to 20% of cases whose cause remains unclear are known as idiopathic RAP. For RAP patients with clear cause, removal of the cause can effectively reduce or prevent recurrence. For patients with idiopathic RAP, the treatment options are not clear and have been subject to debate. At present, the natural course, outcome and therapeutic effect of RAP is still not clear. Therefore, the prospective cohort can clarify the clinical characteristics of RAP more comprehensively and deeply and to accumulate evidence for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent acute pancreatitis.

Exclusion Criteria:

* Unwilling or unable to provide consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients whti recurrent acute pancreatitis come from Changhai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of acute pancreatitis | Through study completion, an average of 1 year
  Acute pancreatitis is diagnosed according to the revised Atlanta classification, which requires 2 of the 3 following criteria: (1) abdominal pain suggestive of pancreatitis, (2) serum amylase and/or lipase greater than 3 times the upper limit of normal, (3) and crosssectional imaging (CT or MRI) findings consistent with acute pancreatitis.

SECONDARY OUTCOMES:
Proportion of patients with different treatment | Through study completion, an average of 1 year
  Treatment mainly contains conservative treatment, surgery, endoscopic intervention, etc. Collect relevant data through medical record.
Characteristics of acute pancreatitis | Through study completion, an average of 1 year
  Collect relevant data through medical record. Characteristics of acute pancreatitis includ etiology, frequency, severity and length of hospital.
Proportion of patients wtih pain in RAP patients | Through study completion, an average of 3 year
  Collect relevant data through pain assessment scales which include severity, frequency, time of duration and other characteristics of pancreatic pain.
Proportion of patients with chronic pancreatitis | Through study completion, an average of 3 year
  Proportion of patients who developed chronic pancreatitis.
Evaluation of quality of life | Through study completion, an average of 3 year
  The level of quality of life in RAP patients is measured using the SF-36.
Evaluation of psychological condition | Through study completion, an average of 3 year
  The psychological condition of RAP patients is measured using DASS-21.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D., Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No